CLINICAL TRIAL: NCT06653426
Title: The Effect of Sodium Butyrate on Menstrual Symptoms in Women
Brief Title: The NaBu Effect on Menstruation in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magdy Milad, MD (Other)
Responsible Party: Sponsor-Investigator, Magdy Milad, MD, Division Chief, MIGS; Medical Director, Center for Complex Gynecology, Northwestern University
Organization: Northwestern University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00220694
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-09

CONDITIONS: Menstrual Symptoms
MeSH Terms: interventions — Butyric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sodium butyrate (NaBu) (Experimental): Participants in the study will be administered Sodium Butyrate (NaBu) in tablet form. Each participant will take a dosage of 2.4 grams, which equates to two tablets, once daily. This regimen will be maintained for a duration of 12 weeks. The supplement is self-administered, and participants are required to record their daily symptom severity in an electronic diary (eDiary) throughout the study period. This intervention aims to assess the effectiveness of NaBu in reducing menstrual symptoms by comparing the average symptom scores during the 12-week treatment period to the baseline scores recorded before starting the supplement.
  Interventions: Dietary Supplement: Sodium Butyrate (NaBu)

INTERVENTIONS:
Dietary Supplement: Sodium Butyrate (NaBu) — Participants will self-administer Sodium Butyrate (NaBu) daily for 12 weeks. The study aims to evaluate the effect of NaBu on menstrual symptoms by comparing symptom severity before and during the intervention. Participants will maintain an electronic diary (eDiary) to record their daily symptom severity, which will be used to assess changes over time. Regular follow-ups will be conducted to monitor progress and address any side effects or concerns.

SUMMARY:
The purpose of this study is to evaluate the effect of once-daily Sodium butyrate (NaBu) on menstrual symptoms in women. The investigators posit that the use of NaBu will reduce menstrual symptoms after taking NaBu for 12 weeks.

DETAILED DESCRIPTION:
The general symptoms of menstruation include abdominal and/or pelvic cramping, lower back pain, bloating, mood swings, and irritability. The exact etiology of these symptoms is not well described. Many pathologies that lead to dysmenorrhea are associated with estrogen-dependent cells, such as endometrial cells, linking estrogen production at the cellular level with symptoms of menstruation.

Sodium butyrate (NaBu) is a food supplement readily available in the US in stores and online. It has been shown to inhibit aromatase, a key enzyme in the estrogen biosynthesis pathway, through a mechanism specific to endometrial cells. The transcription process of estrogen is regulated by up to 10 different promotors, depending on the tissue (Attar, 2006; Simpson, 2002). Aromatase transcription in ovarian endometrioma-derived cells & extra-ovarian endometrioma-derived cells is mediated by Promotor II (Attar 2006). NaBu works by inhibiting the phosphorylation and binding of Activating Transcription Factor 2 (ATF2) to promotor II (Deb, 2006). Thus, NaBu has the potential to reduce estrogen synthesis via the inhibition of the aromatase pathway in cells that use promotor II and in no other tissues.

In this study, the investigators will evaluate the effect of daily NaBu on the baseline symptoms of menstruation in women.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Menstruating regularly or irregularly
* Experiencing menstrual symptoms with an average baseline symptom score of at least 3 on a scale of 0 to 10 for at least one symptom during the initial pre-study rating period.

Exclusion Criteria:

* Pregnant or breastfeeding patient, attempting or anticipating pregnancy.
* Patient with a history of bloating or a sensitive gut (food intolerance) who needs lower fiber levels.
* Patients with known lactose intolerance, other fermentable oligo-, di-, and mono-saccharides, and polyols (FODMAP) intolerances, or small intestinal bacterial overgrowth (SIBO).
* Patients who would require taking daily antacids for the duration of the study.
* Patients with known or suspected chronic hypertension.
* Post-menopausal patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Average Menstrual Symptom Scores | Baseline period (one menstrual cycle before starting NaBu) and the 12-week treatment period.
  The primary outcome measure is the change in average menstrual symptom scores from baseline to the average scores during the 12-week timeframe of taking daily Sodium butyrate (NaBu). Participants will rate their symptoms daily during their menstrual period on a scale of 0 to 10, where 0 indicates no symptoms and 10 indicates the worst possible symptoms (e.g., intolerable pain). The average symptom scores during the 12-week treatment period will be compared to the average baseline score to assess the effectiveness of NaBu in reducing menstrual symptoms. Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy P Milad, MD MS, Principal Investigator — Northwestern Medicine
Locations (1):
- Northwestern University - Northwestern Medicine, Lavin Family Pavilion, Chicago, Illinois, United States

REFERENCES:
- [Background] Tarnowski W, Borycka-Kiciak K, Kiciak A, et al.. Outcome of treatment with butyric acid In irritable bowel syndrome-preliminary report. Gastroenterol Prakt 2013; 1: 43-8
- [Background] Banasiewicz T, Krokowicz L, Stojcev Z, Kaczmarek BF, Kaczmarek E, Maik J, Marciniak R, Krokowicz P, Walkowiak J, Drews M. Microencapsulated sodium butyrate reduces the frequency of abdominal pain in patients with irritable bowel syndrome. Colorectal Dis. 2013 Feb;15(2):204-9. doi: 10.1111/j.1463-1318.2012.03152.x. PMID 22738315
- [Background] Banasiewicz T, Kaczmarek E, Maik J, et al. Quality of life and the clinical symptoms at the patients with irritable bowel syndrome treated complementary with protected sodium butyrate. Gastroenterol Prakt. 2011;5:45-53.
- [Background] Deb S, Zhou J, Amin SA, Imir AG, Yilmaz MB, Lin Z, Bulun SE. A novel role of sodium butyrate in the regulation of cancer-associated aromatase promoters I.3 and II by disrupting a transcriptional complex in breast adipose fibroblasts. J Biol Chem. 2006 Feb 3;281(5):2585-97. doi: 10.1074/jbc.M508498200. Epub 2005 Nov 21. PMID 16303757
- [Background] Zhou J, Gao S, Chen J, Zhao R, Yang X. Maternal sodium butyrate supplement elevates the lipolysis in adipose tissue and leads to lipid accumulation in offspring liver of weaning-age rats. Lipids Health Dis. 2016 Jul 22;15(1):119. doi: 10.1186/s12944-016-0289-1. PMID 27449927
- [Background] Borycka-Kiciak K, Banasiewicz T, Rydzewska G. Butyric acid - a well-known molecule revisited. Prz Gastroenterol. 2017;12(2):83-89. doi: 10.5114/pg.2017.68342. Epub 2017 Jun 13. PMID 28702095
- [Background] Zaleski A, Banaszkiewicz A, Walkowiak J. Butyric acid in irritable bowel syndrome. Prz Gastroenterol. 2013;8(6):350-3. doi: 10.5114/pg.2013.39917. Epub 2013 Dec 30. PMID 24868283
- [Background] Simpson ER, Clyne C, Rubin G, Boon WC, Robertson K, Britt K, Speed C, Jones M. Aromatase--a brief overview. Annu Rev Physiol. 2002;64:93-127. doi: 10.1146/annurev.physiol.64.081601.142703. PMID 11826265
- [Background] Attar E, Bulun SE. Aromatase and other steroidogenic genes in endometriosis: translational aspects. Hum Reprod Update. 2006 Jan-Feb;12(1):49-56. doi: 10.1093/humupd/dmi034. Epub 2005 Aug 25. PMID 16123052